CLINICAL TRIAL: NCT06954584
Title: An Open-label, Randomized Controlled, Multicenter Study With Dual HRD-positive/Negative Cohorts Evaluating Fluzoparib Monotherapy Versus Combination Therapy With Bevacizumab or Dietary Intervention as Maintenance Treatment Following First-line Platinum-based Chemotherapy in Advanced Ovarian Cancer
Brief Title: Fluzoparib+Bevacizumab/Dietary Intervention vs Fluzoparib Monotherapy as First-line Maintenance in HRD+/- Advanced Ovarian Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qinglei Gao, chief physician, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-OC-III-013
Record Dates: First submitted 2025-04-13; First posted 2025-05-01 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HRD-Positive Cohort (Experimental Group): Fluzoparib + Bevacizumab (Experimental): Fluzoparib Capsules : 150 mg orally twice daily (bid) (50 mg/capsule, 3 capsules/dose) .
  Bevacizumab : 15 mg/kg intravenously every 3 weeks until disease progression or intolerable toxicity, with a maximum duration of 15 months .
  Interventions: Drug: Bevacizumab; Drug: Fluzoparib Monotherapy
- HRD-Positive Cohort (Control Group): Fluzoparib Monotherapy (Active Comparator): Fluzoparib Capsules : 150 mg orally bid (50 mg/capsule, 3 capsules/dose)
  Interventions: Drug: Fluzoparib Monotherapy
- HRD-Negative Cohort (Experimental Group 1): Fluzoparib + Dietary Intervention (Experimental): Fluzoparib Capsules : 150 mg orally bid (50 mg/capsule, 3 capsules/dose)
  Interventions: Drug: Fluzoparib Monotherapy; Behavioral: Dietary Intervention
- HRD-Negative Cohort (Experimental Group 2): Fluzoparib Monotherapy (Experimental): Fluzoparib Capsules : 150 mg orally bid (50 mg/capsule, 3 capsules/dose)
  Interventions: Drug: Fluzoparib Monotherapy

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab : 15 mg/kg intravenously every 3 weeks until disease progression or intolerable toxicity, with a maximum duration of 15 months
  Arms: HRD-Positive Cohort (Experimental Group): Fluzoparib + Bevacizumab
Drug: Fluzoparib Monotherapy — 150 mg orally bid (50 mg/capsule, 3 capsules/dose)
Behavioral: Dietary Intervention — Control carbohydrate intake in the daily diet
  Arms: HRD-Negative Cohort (Experimental Group 1): Fluzoparib + Dietary Intervention

SUMMARY:
Fluzoparib has been approved for the first-line maintenance treatment of advanced ovarian cancer in the full population . Previous studies have demonstrated that anti-angiogenic agents enhance tumor cell sensitivity to PARP inhibitors . In vitro evidence suggests that low-carbohydrate culture conditions may restore PARP inhibitor sensitivity in HRD-negative tumor cells. This study aims to validate the survival benefits of fluzoparib combined with bevacizumab in HRD-positive ovarian cancer patients during first-line maintenance therapy and explore the efficacy of fluzoparib combined with a dietary intervention in HRD-negative populations.

ELIGIBILITY:
Inclusion Criteria:

1. The participant voluntarily joins the study, provides written informed consent, demonstrates good compliance, and agrees to follow-up.
2. Female, age ≥18 years (calculated on the day of signing the informed consent form).
3. Histologically confirmed high-grade serous ovarian cancer, fallopian tube cancer, or primary peritoneal cancer ; endometrioid adenocarcinoma of the ovary (grade ≥II) :

   For mixed tumors: The high-grade serous or grade ≥II endometrioid component must exceed 50% .
4. FIGO 2018 staging as Stage III or IV .
5. Documented HRD (Homologous Recombination Deficiency) test results .
6. Completed platinum-based chemotherapy with the following requirements:

   * Patients unable to tolerate chemotherapy for definitive reasons must complete at least 4 cycles of platinum-based chemotherapy .
   * Patients undergoing interval debulking surgery must complete at least 3 cycles of platinum-based chemotherapy post-surgery .
7. Prior to randomization, patients must have no evidence of disease (NED) or achieve complete response (CR) or partial response (PR) after first-line platinum-based chemotherapy, with response maintained until study treatment initiation. Randomization and treatment must begin within 8 weeks after the last chemotherapy dose .

   -CR definition : No radiologic evidence of disease and CA125 ≤ upper limit of normal (ULN).

   -PR definition : ≥30% reduction in tumor size compared to pre-chemotherapy or CA125 reduction ≥90% from baseline (if imaging shows no lesions but CA125 remains above ULN).

   -For patients achieving NED after initial debulking surgery:CA125 must decrease to <1×ULN during treatment and remain <1×ULN within 7 days prior to randomization; or CA125 reduction ≥90% from baseline and no >10% increase within 7 days prior to randomization.

   -Prohibited during/after platinum-based chemotherapy : Concurrent use of other investigational drugs (except endocrine therapy) or treatments.

   -Permitted during chemotherapy : Bevacizumab combination therapy.
8. ECOG Performance Status (PS) : 0-1.
9. Adequate organ function (no blood transfusions or growth factors within 14 days prior to randomization):

   -Absolute neutrophil count (ANC) ≥1.5×10⁹/L.

   -Platelets ≥90×10⁹/L.

   -Hemoglobin ≥9 g/dL.

   -Serum albumin ≥3 g/dL.

   -Total bilirubin ≤1.5×ULN.

   -ALT and AST ≤2.5×ULN.
   * Serum creatinine ≤1.5×ULN.

     1 0.For women of childbearing potential :
   * Negative serum pregnancy test within 72 hours prior to randomization.
   * Agreement to use medically approved contraception during treatment and for 6 months after the last dose .
   * Non-lactating.

   Additional Inclusion Criteria for HRD-Negative Cohort Only :

11. Baseline body mass index (BMI) ≥18.5 kg/m² (BMI = weight [kg]/height [m]²).

Exclusion Criteria:

1. History of other untreated or active malignancies within 5 years (except cured thyroid cancer, basal cell carcinoma, cervical carcinoma in situ, or breast cancer with >3 years of recurrence-free survival after radical surgery).
2. Untreated central nervous system (CNS) metastases :

   -Patients with stable CNS metastases (confirmed by imaging for ≥1 month) after prior systemic/local therapy (e.g., surgery/radiotherapy) and off steroids (>10 mg/day prednisone equivalent) for >2 weeks may be eligible.
3. Prior use of PARP inhibitors (e.g., olaparib, niraparib, rucaparib, pamiparib, fluzoparib).

4 .Inability to swallow tablets or gastrointestinal dysfunction affecting drug absorption (per investigator judgment).

5.Bowel obstruction or gastrointestinal perforation within 3 months prior to randomization.

6.Symptomatic malignant ascites/pleural effusion requiring drainage or drainage within 3 months prior to randomization.

7.Poorly controlled cardiac disease :

* NYHA Class ≥II heart failure.
* Unstable angina.
* Myocardial infarction within 1 year.
* Clinically significant arrhythmias requiring treatment.
* QTc interval >470 ms. 8.Coagulation abnormalities :
* INR >1.5 or PT >ULN +4 seconds.
* Bleeding tendency or current use of thrombolytics/anticoagulants (low-dose LMWH or aspirin prophylaxis permitted).

  9.Clinically significant bleeding within 3 months prior to randomization (e.g., gastrointestinal bleeding, hemorrhagic gastric ulcer, vasculitis).
* If baseline fecal occult blood test is positive, retesting is required. Persistent positivity may necessitate endoscopy.

  10.Active ulcers, unhealed wounds, or fractures . 11.Uncontrolled hypertension (systolic ≥140 mmHg or diastolic ≥90 mmHg despite medication).

  1 2.Grade ≥2 bleeding events (per CTCAE v5.0) within 4 weeks prior to randomization.

  13.Active infection or unexplained fever >38.5°C during screening/prior to randomization.

  14.Immunodeficiency or active hepatitis :
* HIV-positive.
* Active HBV (HBsAg+ and HBV DNA ≥500 IU/mL) or HCV (HCV Ab+ and HCV RNA >ULN).

  1 5.Recent anticancer therapy :
* Chemotherapy, radiotherapy, hormonal therapy, or targeted therapy within 4 weeks prior to study treatment (or 5 half-lives for oral targeted agents).
* Residual toxicity from prior therapy >Grade 1 (CTCAE v5.0; alopecia excluded). 16.Arterial/venous thromboembolism within 6 months prior to randomization (e.g., stroke, transient ischemic attack, DVT, pulmonary embolism).

  17.Hereditary/acquired bleeding disorders (e.g., hemophilia, thrombocytopenia).

  18.Planned use of other systemic anticancer therapies during the study. 19.Any condition that, per investigator judgment, may lead to premature study termination.

Additional Exclusion Criteria for HRD-Negative Cohort Only :

20. Unintentional weight loss ≥5% within 3-6 months or presence of cachexia .

21. Nutritional risk :

-NRS2002 score ≥3 or need for nutritional support. 22.Diabetes requiring insulin or insulin secretagogues . 23.Acute liver disease/dysfunction . 24.Active chronic or acute kidney disease/dysfunction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2030-05-01 (Estimated); Study Completion 2032-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 96 months
  The time from randomization to the occurrence of disease progression (as per RECIST v1.1) or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Time to Progression (TTP) | From date of randomization until the date of first documented CA125 progression (as per GCIG-CA125 criteria) or disease progression (as per RECIST criteria), whichever came first, assessed up to 96 months
  The time from randomization to CA125 progression (as per GCIG-CA125 criteria) or disease progression (as per RECIST criteria), whichever occurs first.
Time to Discontinuation or Death (TDT) | From date of randomization until the date of first documented discontinuation of study treatment or death from any cause, whichever came first, assessed up to 96 months
  The time from randomization to discontinuation of study treatment or death from any cause, whichever occurs first.
ime to First Subsequent Therapy (TFST) | From date of randomization until the date of first documented initiation of subsequent anti-tumor therapy for ovarian cancer, or death, assessed up to 96 months
  The time from randomization to the initiation of subsequent anti-tumor therapy for ovarian cancer, or death.
Best Overall Response (BOR) | From date of randomization until disease progression or recurrence, assessed up to 96 months
  The best objective response recorded from randomization until disease progression or recurrence.
Overall Survival (OS) | From date of randomization until the date of death from any cause, assessed up to 96 months
  The time from randomization to death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No